CLINICAL TRIAL: NCT02742480
Title: Dabigatran Study in the Early Phase of Stroke. New Neuroimaging Markers and Biomarkers Study (SEDMAN STUDY)
Acronym: SEDMAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: JKB-DAB-2016-01
Record Dates: First submitted 2016-04-08; First posted 2016-04-19 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Cardioembolic Stroke
Keywords: stroke; oral anticoagulants; cardioembolic
MeSH Terms: conditions — Embolic Stroke; Stroke | interventions — Dabigatran; Acenocoumarol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Dabigatran: 300 patients treated with dabigatran under the habitual clinical practice.
  Interventions: Drug: Dabigatran
- Acenocoumarol: 200 patients treated with acenocoumarol under the habitual clinical practice.
  Interventions: Drug: Acenocoumarol

INTERVENTIONS:
Drug: Dabigatran
  Groups: Dabigatran
Drug: Acenocoumarol
  Groups: Acenocoumarol

SUMMARY:
SEDMAN study is a prospective multicenter investigator initiated study (IIS). The main idea is to look by Genome Wide Association (arrays that determine more than 1 million polymorphisms) genetic risk factors associated with response to dabigatran. To conduct the study, the goal is to recruit 300 patients with ischemic stroke with cardioembolic etiology treated with dabigatran and 200 treated with Acenocoumarol to determine if genetic risk factors are associated with the occurrence of any bleeding or vascular event in a year follow-up.

DETAILED DESCRIPTION:
Data will be analyzed through GWAS analysis. The results will be analyzed by experienced genotypic bioinformatics: Plink, Haploview, STATA, IMPUTE2, SNPtest, GTOOL, Galaxy management. In addition, the investigators have support of Spanish Consortium for Genetics of Stroke (Genestroke). The PLINK software is the main program for the analysis of GWAS. Using this software we can clean the raw results of genotyping platforms and determine the presence of risk alleles associated with resistance to the study drugs. Haploview software will be used for data management and graphics for significance analysis. STATA statistical software is a data management and very useful for the creation of Q_Q plots graphs that assist in the interpretation of genotypic results. GTOOL, SNPtest and IMPUTE2 are software for data imputation and analysis of imputed data through the information available in the 1000 Genomes Project.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes who are ≥ 18 years of age
* Patients with stroke or TIA in last 14 days and a diagnosis of non-valvular atrial fibrillation who initiate treatment with dabigatran or classical ACOs (acenocoumarol) to prevent stroke or non-CNS systemic embolism.
* Patients with mild/moderate strokes (i.e. strokes less than 2/3 of vascular territory with initial ASPECTS on first CT/MRI > 6 and NIHSS <25).
* Patients who have an overall condition which allow the 12 months' follow-up.

Exclusion Criteria:

* Patients with an indication of oral anticoagulants for primary prevention or with an indication other than cardioembolic etiology.
* Patients with contraindications to use anticoagulants.
* Patients who do not wish to participate in the study and have not signed informed consent.
* Patients with non-controlled hypertension or hypertensive crisis will be also excluded.
* Patients with a life expectancy of less than one year.
* Patients with psychological or social factor which not allow a correct follow-up.
* Patients with severe/disabling strokes (i.e. more than 2/3 of vascular territory, NIHSS≥25).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes who are at least 18 years of age with a diagnosis of non-valvular atrial fibrillation and stroke or TIA and after taking the decision to perform pharmacological prophylaxis with dabigatran or acenocoumarol under the approved indication and the recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-06-28 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Stroke (including TIA) or systemic embolism (Efficacy) | 1 year
  Efficacy will be defined as stroke (including TIA) or systemic embolism
Any type of hemorrhage (clinically minor and major bleeding) | 1 year
  Safety variable will include any type of hemorrhage (clinically minor and major bleeding).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain